CLINICAL TRIAL: NCT00588640
Title: A Phase I/II Study of D-Methadone in Patients With Chronic Pain
Brief Title: Study of D-Methadone in Patients With Chronic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01-017
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-06

CONDITIONS: Pain; Bladder Cancer; Breast Cancer; CNS Cancer; Colon Cancer; Esophageal Cancer; Pancreatic Cancer; Prostate Cancer; Uterine Cancer; Head and Neck Cancer; Eye Cancer; Otorhinolaryngologic Neoplasms
Keywords: Pain; HEENT cancer
MeSH Terms: conditions — Pain; Urinary Bladder Neoplasms; Breast Neoplasms; Central Nervous System Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Uterine Neoplasms; Head and Neck Neoplasms; Eye Neoplasms; Otorhinolaryngologic Neoplasms | interventions — D-methadone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Phase I, Group (Experimental): This is an open label dose-ranging trial. The first cohort of 8 patients will receive 40mg of d-methadone every 12 hours.
  Interventions: Drug: d-Methadone
- Phase II, Group I (Experimental): patients receiving around the clock opioid therapy-No patients were accrued to this group
  Interventions: Drug: D-methadone
- Phase II, Group II (Experimental): patients not receiving around the clock opioid therapy.No patients were accrued to this group
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: d-Methadone — 8 subjects to receive 40 mg d-Methadone twice a day
  Arms: Phase I, Group
Drug: D-methadone — After randomization, patients will take the study drug or placebo for 12 days and then they will cross-over to the opposite arm for another 12 days. The study will end on day 24.
  Arms: Phase II, Group I
Drug: placebo — After randomization, patients will take the study drug or placebo for 12 days and then they will cross-over to the opposite arm for another 12 days. The study will end on day 24.
  Arms: Phase II, Group II

SUMMARY:
The purpose of this study is to determine the safest dose of d-methadone that can be given, without causing severe side effects in most patients with chronic pain. Patients are being asked to participate in the Phase I portion of this study.

ELIGIBILITY:
Inclusion Criteria:

Phase I and Phase II portions of the study:

* 18 years of age or older
* Chronic pain with average 24 hour intensity rated at least 3 on a verbal numerical scale from 0-10 during the 24 hours prior to study entry.
* Give informed consent to participate in this study.
* Karnofsky Performance Score (KPS) >= to 80
* Negative urine pregnancy test, verified by the study nurse, at study entry (for women of child-bearing potential). Patients must also use a medically approved contraceptive method during the study period.

Phase I only:

* Responsible companion living with patient during study.

Phase II only:

* Group 1 -- Patients must be taking chronic opioid therapy (long acting morphine, long acting oxycodone, transdermal fentanyl) at a stable dose for a minimum of four days. The dose of as needed short acting opioid does not need to be stable.
* Group 2 -- Patients must not be receiving opioids and must have cancer related neuropathic pain secondary to post-chemotherapy peripheral neuropathy, post-radiation and/or post surgical plexopathy, radiculopathy or neuropathy, or post- herpetic neuralgia.

Exclusion Criteria:

Phase I and Phase II:

* Known hypersensitivity to methadone
* Patient taking methadone or with a history of methadone treatment within one month of study enrollment.
* Patient that requires changes in the dose of one of the following medications within 2 weeks of study enrollment:

  * Abacavir,
  * Benzodiazepines,
  * Carbamazepine,
  * Efavirenz,
  * Fluconazole,
  * Fluvoxamine,
  * FOS amprenavir,
  * Fosphenytoin,
  * Naltrexone,
  * Nelfinavir,
  * Nevirapine,
  * Phenytoin,
  * Rifampin,
  * Rifapentine,
  * Risperidone,
  * Ritonavir,
  * St. John's Wort,
  * Zidovudine
* Hepatic function tests (SGOT, alkaline phosphatase, bilirubin) greater than 2 times the upper limit of normal or creatinine greater than 1.4 within 30 days of study entry.
* Neurologic or psychiatric disease sufficient, in the investigator's opinion, to compromise data collection.
* Women who are pregnant or nursing.
* Women of childbearing potential who do not agree to use a medically recognized method of contraception during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Moryl, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving D-methadone 40 mg: Patient Receiving D-methadone 40 mg
Period: Overall Study
Arm/Group | Patients Receiving D-methadone 40 mg
Started | 10
Completed | 8
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Ineligible Patient | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients Receiving D-methadone 40 mg
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number Who Reached a Safe Dose
Description: The number of patients who reached a safe and well tolerated dose of d-methadone
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Phase I, Cohort l: oral d-methadone 40 mg
  d-Methadone: 8 subjects to receive 40 mg d-Methadone twice a day
Arm/Group | Phase I, Cohort l
Number analyzed (Participants) | 8
participants | 8

ADVERSE EVENTS:
Arm/Group | Patients Receiving D-methadone 40 mg
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving D-methadone 40 mg (N=9)
Pain - Neck (General disorders) | 1 (1)
Pain - Back (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving D-methadone 40 mg (N=9)
Constipation (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Glucose, high (hyperglycemia) (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Pain - Joint (General disorders) | 1 (1)
Pain - Pain NOS (General disorders) | 1 (1)
Prolonged QTc interval (Cardiac disorders) | 3 (3)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes